CLINICAL TRIAL: NCT03135704
Title: Comparison of Two Treatments for Low Back Pain: "Re Spine" vs. Physiotherapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HYMC-0025-17
Record Dates: First submitted 2017-04-20; First posted 2017-05-01 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "Re Spine" Mattress (Active Comparator): Adults suffering low back pain will treat their low back pain using the "Re Spine" mattress
  Interventions: Device: "Re Spine"
- Physiotherapy (Active Comparator): Adults suffering low back pain will treat their low back pain using conventional physiotherapy protocols
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Device: "Re Spine" — A new mattress design made of special materials and built in a specially shaped structure that allows the brain to relax the body and dissipate tension accumulated on the lumbar spine.
  Arms: "Re Spine" Mattress
Other: Physiotherapy — Usual protocol for treatment of low back pain
  Arms: Physiotherapy

SUMMARY:
The objective of this study is to assess the effectiveness of the "Re Spine" mattress, which was designed as an alternative to physiotherapy in the treatment of low back pain (LBP).

ELIGIBILITY:
Inclusion Criteria:

* Low back pain

Exclusion Criteria:

* None

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in low back pain | 1 day, 6 weeks, 3 months
  Pain levels will be measured using the Visual Analogue Scale (VAS) on the first day of study and 6 weeks, and 3 months after treatment at end of study.
Effectiveness of treatment | 1 day, 6 weeks, 3 months
  Effectiveness of treatment will be assessed based on Oswestry Disability Index and Mini Sleep Questionnaire on the first day of study and 6 weeks, and 3 months after treatment at end of study.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Behrbalk, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe Medical Center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No